CLINICAL TRIAL: NCT04907149
Title: A Phase 1, Open-label Study to Investigate the Pharmacokinetics and Metabolism of GLPG3970 in Healthy Male Subjects Following a Single Oral Dose of GLPG3970 Relative to an Intravenous [14C]GLPG3970 Microtracer and Single Oral [14C]GLPG3970 Administration
Brief Title: Evaluation of Mass Balance and Absolute Bioavailability of GLPG3970
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG3970-CL-107; 2021-000711-23 (EudraCT Number)
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absolute Bioavailability - Period 1 (Experimental): Participants will receive GLPG3970 under fasted conditions followed by an intravenous (i.v.) microtracer microdose of [14C]GLPG3970 on Day 1.
  Interventions: Drug: GLPG3970 film-coated tablet; Drug: [14C]GLPG3970 solution for infusion
- Mass Balance - Period 2 (Experimental): Participants will receive [14C]GLPG397 under fasted conditions on Day 1.
  Interventions: Drug: [14]GLPG3970 oral solution

INTERVENTIONS:
Drug: GLPG3970 film-coated tablet — Participants will receive a single oral dose of GLPG3970.
  Arms: Absolute Bioavailability - Period 1
Drug: [14C]GLPG3970 solution for infusion — Participants will receive an i.v. microtracer microdose.
  Arms: Absolute Bioavailability - Period 1
Drug: [14]GLPG3970 oral solution — Participants will receive a single oral dose [14C]GLPG3970.
  Arms: Mass Balance - Period 2

SUMMARY:
A study in healthy male volunteers to assess how the radiolabelled test medicine is taken up and broken down by the body when given by short infusion into a vein and when given by the mouth in the form of a tablet and an oral solution.

ELIGIBILITY:
Inclusion Criteria:

* Male between 30 and 64 years of age (extremes included), on the date of signing the informed consent form (ICF).
* A body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
* Having a regular (at least) daily defecation pattern (i.e. 1 to 3 times per day).

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Participant has participated in a [14C]radiolabeled study within the past 12 months.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 month or 10 mSv in the last 5 years. Occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017 (UK, 2017), cannot participate in the study.

This list only contains the key exclusion criteria.

Ages: 30 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F [%]) of GLPG3970 | From Day 1 pre-dose until Day 4 in Period 1
Recovery of total radioactivity excreted in urine expressed as a percentage of the administered dose (Ae%). | From Day 1 pre-dose until Day 8 in Period 2
Recovery of total radioactivity excreted in feces expressed as a percentage of the administered dose (Ae%). | From Day 1 pre-dose until Day 8 in Period 2

SECONDARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations. | From Day 1 through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Tankisheva, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No